CLINICAL TRIAL: NCT03138590
Title: Investigating Accelerated Learning in Healthy Subjects
Brief Title: Investigating Accelerated Learning in Healthy Subjects: Trigeminal Nerve Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No relevant anymore
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-34 TN
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Healthy Adults
Keywords: transcranial Direct Current Stimulation (tDCS); accelerate learning; memory

STUDY DESIGN:
Intervention Model Description: participants will be randomly assigned to one of 2 groups: (1) active tDCS (2) sham tDCS
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (Experimental): Active transcranial Direct Current Stimulation targeting the trigeminal nerve
  Interventions: Device: Transcranial Direct Current Stimulation- Neuroconn DC Stimulator PLUS
- Sham tDCS (Sham Comparator): Sham transcranial Direct Current Stimulation targeting the trigeminal nerve
  Interventions: Device: Transcranial Direct Current Stimulation- Neuroconn DC Stimulator PLUS

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation- Neuroconn DC Stimulator PLUS — Transcranial Direct Current Stimulation targeting the trigeminal nerve

SUMMARY:
The purpose of this study is to investigate whether it is possible to accelerate learning and improve associative memory performance in healthy subjects, by applying transcranial Direct Current Stimulation (tDCS) targeting the trigeminal nerve during a verbal paired-associate learning task

DETAILED DESCRIPTION:
Associative memory refers to remembering the association between two items, such as a face and a name or a word in English and the same word in another language. It is not only important for learning, but it is also one of the first aspects of memory performance that is impacted by aging and by Alzheimer׳s disease. For decades, neuroscientists have investigated associative learning and memory and ways to accelerate and enhance associative learning and memory.

Transcranial Direct Current stimulation (tDCS) is a non-invasive and painless electrical stimulation technique that has demonstrated to accelerate learning and improve memory in some studies. To investigate whether it is possible to accelerate learning and improve associative memory using tDCS, the performance in a Verbal Paired-Associate memory task of 2 groups will be compared. The first group will get active tDCS during the verbal paired-associate learning task. The second group will get sham tDCS during the verbal paired-associate learning task.

ELIGIBILITY:
Inclusion Criteria:

* Native English Speaker

Exclusion Criteria:

* History of severe head injuries, epileptic insults, or heart disease.
* Severe psychiatric disorders and severe untreated medical problems
* Acquainted with the foreign language used in the learning task
* Contraindications for tDCS (e.g. pregnant, implanted devices)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas of Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (4.67) | 21.1 (2.33) | 21.3 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
Beck Depression Inventory Scale [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Measure Description: The Beck Depression Inventory (BDI, BDI-1A, BDI-II), created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.
  The Beck Depression Inventory uses the following scale to assess patients: 0 - 13: Minimal depression, 14 - 19: Mild depression, 20 - 28: Moderate depression, 29 - 63: Severe depression Min score: 0; Max Score: 63; The higher the score the more mood
  units on a scale | 5 (5.65) | 4.3 (4.34) | 4.65 (4.92)
Beck Anxiety Inventory Scale [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Measure Description: The Beck Anxiety Inventory (BAI), created by Aaron T. Beck and other colleagues, is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults.
  The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are:
  0-7: minimal anxiety 8-15: mild anxiety 16-25: moderate anxiety 26-63: severe anxiety
  units on a scale | 2.6 (2.07) | 2.6 (2.99) | 2.6 (2.5)
Mini Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Measure Description: The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
  Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
  units on a scale | 29.3 (1.06) | 29.5 (0.972) | 29.4 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: Associative Memory Assessed by a Verbal Paired-Associate Test
Description: Changes in performance in the Verbal Paired-Associate memory task is compared between the 2 groups (1. Active tDCS 2. Sham tDCS) to investigate the influence of tDCS on Associative Memory.
Time Frame: 1 week after stimualtion
Measure: Mean (Standard Deviation); unit: percentage of words recalled from V1
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 10 | 10
percentage of words recalled from V1 | 32.9 (16.2) | 38.1 (18.6)

ADVERSE EVENTS:
Time Frame: One Week
Description: Before the end of the experiment, participants were asked to fill out a questionnaire (Brunoni et al., 2011) to assess their experiences of possible side effects (e.g., headache, neck pain, and scalp pain) related to the stimulation on a 4-point scale (1 = absent, 2 = mild, 3 = moderate, and 4 = severe).
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol: Protocol 17-34 TN (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03138590/Prot_001.pdf